CLINICAL TRIAL: NCT00013364
Title: Effects of Stimulus Validity on Speech Recognition
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: C1850R
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Hearing Impaired
Keywords: Hearing loss, speech recognition
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Talker variability

SUMMARY:
The effects of talker variability will be investigated with four groups of listeners (young normal-hearing; old normal-hearing; young hearing-impaired; old hearing-impaired). Experimental conditions will include between-talker differences, speaking rate, lexical difficult and semantic/linguistic context. A preliminary experiment will evaluate the relative merit of adaptive vs fixed-level methods of stimulus presentation.

ELIGIBILITY:
Hearing impaired

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 1998-04; Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D., Program Analyst — Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Nancy Roceleau, Program Analyst — Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, West Los Angeles, Los Angeles, California, United States